CLINICAL TRIAL: NCT07125105
Title: Integrating Art Therapy and Adapted Physical Activity: Toward Improved Quality of Life in Patients With Myasthenia Gravis
Acronym: APART-MG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universite du Littoral Cote d'Opale (Other)
Collaborators: University Hospital, Lille (Other); Fondation Maladies Rares (French Foundation for Rare Diseases) (Unknown); AFM Téléthon (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-A00781-48; 15522 (Other: Fondation Maladies Rares)
Record Dates: First submitted 2025-07-06; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia Gravis; Art Therapy; Adapted Physical Activity; Randomized; Rare Neuromuscular Diseases; Crossover Trial; Quality of Life; Psychosocial Intervention; Fatigue in Chronic Illness; Mental Health in Rare Diseases; Non-pharmacological Interventions; Dramatherapy
MeSH Terms: conditions — Myasthenia Gravis | interventions — Art Therapy; Psychodrama

STUDY DESIGN:
Intervention Model Description: This is a two-arm crossover trial. Participants will be randomly assigned to one of two sequences: (1) Adapted Physical Activity (APA) followed by APA combined with Art Therapy (AT), or (2) APA + AT followed by APA alone. Each intervention phase consists of 10 sessions over 6 weeks, separated by a 46-week washout period to minimize carryover effects.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, participants and care providers will not be blinded to group allocation. However, outcome assessments will be conducted by an independent evaluator who is blinded to the intervention sequence in order to minimize assessment bias. This includes the administration and interpretation of physical performance tests and questionnaires at all evaluation timepoints.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted Physical Activity Only (Experimental): Participants receive 10 individualized sessions of adapted physical activity (45-60 minutes each), designed according to neuromuscular rehabilitation guidelines. The sessions focus on strength, endurance, and movement awareness, and are tailored to the physical limitations and fatigue patterns typical of patients with Myasthenia Gravis . No artistic or expressive components are included
  Interventions: Behavioral: Adapted Physical Activity Only
- Adapted Physical Activity + Art Therapy (Experimental): Participants receive 10 individualized sessions of adapted physical activity (45-60 minutes each) incorporating expressive and artistic components inspired by movement-based art therapy (e.g., dramatization, role-play, symbolic movement). These integrated sessions aim to enhance physical engagement while also addressing emotional expression, body image, and psychosocial well-being. The approach is co-constructed with the participant based on a preliminary qualitative assessment.
  This intervention combines adapted physical activity with movement-based art therapy techniques. The art therapy component is not administered separately but is fully integrated into the APA sessions, forming a unified intervention model. Exercises include expressive movement, dramatization, and body awareness activities delivered by APA specialists with complementary training in art-based methods.
  Interventions: Behavioral: Adapted Physical Activity + Art Therapy

INTERVENTIONS:
Behavioral: Adapted Physical Activity Only — This intervention consists of 10 individual Adapted Physical Activity (APA) sessions over five weeks, each lasting 45 to 60 minutes. Sessions are delivered by a trained APA instructor and focus on muscle strengthening, endurance, and body awareness. Exercises are tailored to the functional capacities and fatigability of patients living with Myasthenia Gravis. The delivery format includes a mix of in-person and remote sessions, with individualized adaptation based on patient needs.
  Other Names: Standard APA sessions
  Arms: Adapted Physical Activity Only
Behavioral: Adapted Physical Activity + Art Therapy — This intervention includes 10 individualized sessions of APA integrated with movement-based Art Therapy, delivered over five weeks (45-60 minutes each). The program incorporates creative and expressive methods (e.g., role play, improvisation, dramatized movement, dramatherapy) within a therapeutic physical activity framework. It is designed to support both physical functioning and psychosocial well-being. The artistic dimension is adapted to the patients' preferences and capacities, as identified during the baseline anamnesis interview.
  Other Names: Artistic APA; Movement-based expressive APA; Dramatherapy
  Arms: Adapted Physical Activity + Art Therapy

SUMMARY:
Myasthenia Gravis (MG) is a rare neuromuscular disease characterized by fluctuating muscle weakness and excessive fatigability. Although medical treatments have improved, MG continues to significantly impact patients' physical, emotional, and social well-being. Current care primarily focuses on symptom management, often overlooking the broader psychosocial needs of patients.

This study explores an innovative and holistic approach combining Adapted Physical Activity (APA) and Art Therapy (AT) to improve quality of life in adults with MG. The intervention includes two 6-week phases in a crossover design: one with APA alone and one combining APA with personalized AT sessions focused on body awareness, movement, and creative expression.

The investigators hypothesize that the addition of AT to a standardized APA program will significantly enhance patients' engagement and well-being, resulting in improved quality of life, reduced fatigue, and better mental health outcomes.

A total of 102 adult participants will be recruited from several hospitals in northern France (Lille, Dunkerque, Calais, Boulogne-sur-Mer, and Saint-Omer). Participants will be randomly assigned to begin with either APA alone or APA+AT. All interventions are tailored to the specific needs of MG patients and will be delivered both in person and online, depending on participant needs.

Outcomes will be evaluated using standardized questionnaires (e.g., MG-QOL15, FSS, HADS), physical performance tests (e.g., handgrip strength, sit-to-stand), and accelerometry. Qualitative data will be collected through semi-structured interviews, ethnographic observations and art based research to better understand patients' experiences.

The study has received ethical approval from the French National Ethics Committee (CPP) and involves minimal risk. Participation is voluntary, with no financial compensation. This protocol may pave the way for broader application of APA+AT models in other rare or chronic conditions that involve fluctuating fatigue and psychosocial complexity.

DETAILED DESCRIPTION:
This study investigates the feasibility and impact of a combined Adapted Physical Activity (APA) and movement-based Art Therapy (AT) intervention for adults living with Myasthenia Gravis (MG). MG is a rare autoimmune disorder affecting neuromuscular transmission, often leading to fluctuating muscle weakness and fatigue. Despite medical advances, MG continues to significantly impact patients' psychosocial well-being and functional autonomy.

Growing evidence supports the use of APA and psychosocial therapies to improve outcomes in chronic neurological conditions. However, no interventional study to date has tested the integration of APA and AT in the MG population. This research protocol addresses this gap by evaluating a crossover intervention comparing two 5-week programs: one involving APA only, and one integrating APA with AT.

The study is a monocentric, randomized crossover trial including 102 adult participants recruited from neurology departments in northern France. Each participant will complete both interventions in randomized order, separated by a 46-week washout period. Stratified randomization will be applied based on sex, age, and MG-ADL score.

The AT component will include movement-based techniques (e.g., dramatization, expressive motion), tailored to each participant's capacity and familiarity with artistic expression. Pre-intervention interviews will guide the personalization of the AT sessions. The primary outcome is change in quality of life (MG-QOL15) at 3-month follow-up. Secondary outcomes include fatigue, anxiety/depression, physical activity, and physical function measures. A qualitative dimension using semi-structured interviews and ethnographic observations will provide insight into patient experiences and psychosocial responses.

This study is designed as a minimal risk interventional trial (RIPH2), with ethical approval granted by the Comité de Protection des Personnes (CPP) and compliance with CNIL data protection standards.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of myasthenia gravis of any form established by a referring neurologist.
* Patients followed at Lille University Hospital and its partners (Neuromuscular Diseases Reference Center, hospitals of the Côte d'Opale, home care services), or at Amiens University Hospital.
* No major contraindications to participating in adapted physical activity and/or art therapy, as evaluated by the medical team.
* Availability to attend all 10 sessions of the APA-only program and the combined APA + AT program, according to the cross-over design.
* Signed informed consent after being informed about the objectives and requirements of the project.

Exclusion Criteria:

* Severe comorbidities limiting participation in adapted physical activity or art therapy.
* Advanced cognitive decline or severe neuropsychiatric disorders preventing understanding and participation.
* Unstable medical treatment with recent changes that may affect fatigability or physical capacity / poorly controlled myasthenia gravis.
* Physical inability to participate in adapted physical activity or art therapy, even with adaptations.
* Unavailability to complete the entire protocol (e.g., relocation, prolonged absence).
* Refusal or inability to provide informed consent (e.g., patient under guardianship without legal authorization).
* Difficulty accessing the intervention locations without possible alternatives such as remote or home-based sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life (MG-QOL15) | 3 and 6 months post-intervention
  Change in quality of life will be assessed using the Myasthenia Gravis Quality of Life 15-item questionnaire (MG-QOL15), a validated tool measuring the impact of MG on patients' physical, psychological, and social well-being. The total score ranges from 0 to 60, with higher scores indicating greater impairment. The main comparison will be between APA alone and APA + AT phases.

SECONDARY OUTCOMES:
Change in Fatigue Severity (FSS) | 3 and 6 months post-intervention
  Fatigue will be assessed using the Fatigue Severity Scale (FSS), a 9-item self-report questionnaire evaluating perceived fatigue and its impact on daily functioning. Higher scores indicate more severe fatigue. The comparison will be made between APA and APA+AT phases.
Change in Anxiety and Depression (HADS) | 3 and 6 months post-intervention
  Emotional status will be assessed using the Hospital Anxiety and Depression Scale (HADS), a validated 14-item questionnaire with two subscales measuring anxiety and depression. Higher scores reflect higher psychological distress. Effects of both intervention phases will be compared.
Change in Physical Activity Level (IPAQ + Accelerometry) | 3 and 6 months post-intervention
  Physical activity will be measured using the International Physical Activity Questionnaire (IPAQ, short form) and intermittent use of accelerometers (ActiGraph wGT3X-BT) to provide both subjective and objective measures of physical activity intensity and duration.
Change in Activities of Daily Living (MG-ADL) | 3 and 6 months post-intervention
  Functional autonomy will be evaluated using the Myasthenia Gravis Activities of Daily Living (MG-ADL) scale, an 8-item instrument assessing the impact of MG on daily functioning. The scale ranges from 0 (no impairment) to 24 (severe impairment).
Change in Handgrip Strength (Takei Dynamometer) | 3 and 6 months post-intervention
  Muscular strength will be assessed using the Handgrip Strength Test with a Takei dynamometer. Participants will perform two trials with each hand, and the best result will be recorded for analysis.
Change in Lower Limb Endurance (30-Second Sit-to-Stand Test) | 3 and 6 months post-intervention
  Lower limb endurance and functional strength will be evaluated using the Sit-to-Stand Test. Participants will be instructed to stand up and sit down from a chair as many times as possible in 30 seconds.
Change in Cardiovascular Endurance (3-Minute Stepper Test) | 3 and 6 months post-intervention
  Cardiovascular endurance will be assessed using a 3-minute adapted stepper test. Heart rate and number of steps will be recorded and compared across timepoints.
Change in Balance (Timed Unipedal Stance Test) | 3 and 6 months post-intervention
  Balance will be measured using the Unipedal Stance Test (UPST). Participants will be asked to stand on one foot with eyes open; the duration they can maintain balance will be recorded.

OTHER OUTCOMES:
Thematic Analysis of Semi-Structured Interviews | Baseline (Day 0), Post-Intervention (Week 6 and Week 58), and Follow-up (Month 3 and Month 6 after each intervention phase)
  Participants will take part in semi-structured interviews to explore their lived experiences of illness, care, and engagement with the intervention. Interviews will be audio-recorded, transcribed, and thematically analyzed to identify psychosocial themes related to coping, self-image, and perceived benefit.
Ethnographic Observations and Field Notes | From Day 0 (Baseline) through study completion, approximately 15 months
  Ethnographic data will be collected through participant observation during intervention sessions, informal interviews, and field notes. Observations will focus on emotional expression, engagement, social interaction, and body language. The material will be analyzed thematically to assess the psychosocial impact of the interventions.
Drawing-Based Creative Expression Analysis | Day 0 (Baseline), immediately post-intervention (Weeks 5 and 56), and follow-up at Month 3 and Month 6 post-intervention
  Drawing activities will be integrated into interviews as creative elicitation tools. Participants will be invited to draw representations of their illness, body image, and emotional states. These drawings will be analyzed visually and thematically to explore symbolic content and changes over time.
Identity Box-Based Narrative Analysis | Day 0 (Baseline), immediately post-intervention (Weeks 5 and 56), and follow-up at Month 3 and Month 6 post-intervention
  Participants will be invited to bring, select or create personal objects to create "identity boxes" as part of the interviews. These objects serve as narrative anchors to facilitate reflection and storytelling. The content and associated narratives will be thematically analyzed to assess psychosocial transformation and meaning-making processes.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Porrovecchio, PhD, Principal Investigator — Université du Littoral Cote d'Opale; Céline Tard, PhD Dr, Principal Investigator — University Hospital of Lille
Locations (1):
- Lille University Hospital, Lille, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No
This study involves rare disease participants and collects sensitive psychosocial and qualitative data. Data will not be shared to ensure participant confidentiality and in accordance with French data protection laws (CNIL/MR001 framework).